CLINICAL TRIAL: NCT00909532
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of VX-770 in Subjects With Cystic Fibrosis and the G551D Mutation
Brief Title: Study of Ivacaftor in Cystic Fibrosis Subjects Aged 12 Years and Older With the G551D Mutation
Acronym: STRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX08-770-102
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Cystic Fibrosis
Keywords: Fibrosis; Pancreatic Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis; Pancreatic Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects who received placebo every 12 hours (q12h) for up to 48 weeks.
  Interventions: Drug: Placebo
- 150 mg Ivacaftor q12h (Experimental): Subjects who received 150 mg of ivacaftor q12h for up to 48 weeks.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor — 150-mg tablets given orally q12h for up to 48 weeks
  Other Names: VX-770
  Arms: 150 mg Ivacaftor q12h
Drug: Placebo — Tablet given orally q12h for up to 48 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of ivacaftor in subjects with cystic fibrosis aged 12 years and older who have the G551D mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. Ivacaftor is a potent and selective CFTR potentiator of wild-type, G551D, F508del, and R117H forms of human CFTR protein. Potentiators are pharmacological agents that increase the chloride ion transport properties of the channel in the presence of cyclic AMP-dependent protein kinase A (PKA) activation.

DETAILED DESCRIPTION:
This was a phase 3 study in subjects with cystic fibrosis (CF) age 12 years and older who have a G551D-CFTR mutation and percent predicted forced expiratory volumn in 1 second (FEV1) between 40% and 90%.

Based on in vitro studies and pharmacologic, pharmacokinetic (PK), and safety profiles, ivacaftor was selected for clinical development as a possible treatment for patients with CF. Patients with the G551D mutation were the targeted population for this study because ivacaftor is a potentiator of the gating function of the CFTR protein, and the most prevalent mutation with a gating defect in CF is the G551D mutation.

This study was designed to further evaluate the efficacy of ivacaftor in subjects with CF who have a G551D-CFTR gene mutation and to evaluate safety in this population over a longer period than previously studied.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis (CF) and G551D mutation in at least 1 allele
* Forced expiratory volume in 1 second (FEV1) of 40% to 90% (inclusive) of predicted normal for age, gender, and height at Screening.
* No clinically significant abnormalities that would have interfered with the study assessments, as judged by the investigator
* Willing to use highly effective birth control methods during the study

Exclusion Criteria:

* History of any illness or condition that might confound the results of the study or pose an additional risk in administering study drug to the subject
* Acute respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks of Day 1 of the study
* History of alcohol, medication or illicit drug abuse within one year prior to Day 1
* Abnormal liver function ≥ 3x the upper limit of normal
* Abnormal renal function at Screening
* History of solid organ or hematological transplantation
* Pregnant, planning a pregnancy, breast-feeding, or unwilling to follow contraception requirements
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within 30 days prior to Screening
* Use of inhaled hypertonic saline treatment
* Concomitant use of any inhibitors or inducers of cytochrome P450 3A4 (CYP 3A4)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie W. Ramsey, MD, Principal Investigator — Children's Hospital and Regional Medical Center, Seattle, Washington, USA; Stuart Elborn, MD, Principal Investigator — Respiratory Medicine Group, Queen's University of Belfast, Belfast, Northern Ireland, UK
Locations (65):
- United States (39):
  - University of Alabama, Birmingham, Alabama
  - Kaiser Permanente Medical Care Program, Oakland, California
  - Cystic Fibrosis Research Office, Stanford University, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Emory Cystic Fibrosis Center, Atlanta, Georgia
  - St. Luke's CF Clinic, Boise, Idaho
  - Children's Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Pulmonary, Allergy & Critical Care Medicine, University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Adult Pulmonary/ CF, University of Nebraska Medical Center, Omaha, Nebraska
  - Monmouth Medical Center, Long Branch, New Jersey
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Pediatric & Pulmonary Division, Rainbow Babies/Case Western, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Division of Pulmonary and CCM, University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - The Children's Hospital Westmead, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Children's Hospital Brisbane, Herston, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - Lung Institute of Western Australia, Nedlands, Western Australia
  - Princess Margaret Hospital for Children, Subiaco, Western Australia
- Canada (4):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - CF Center, Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital - MUHC, Montreal, Quebec
- FN Motol, Prague, Czechia
- France (3):
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - Centre de Perharidy, Roscoff
- Germany (4):
  - Kinder- und Jugendklinik Universitätsklinikum Erlangen, Erlangen
  - Mukoviszidose-Zentrum am Klinikum der Friedrich-Schiller-Universität Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - Klinikum der LMU München, Dr. von Haunersches Kinderspital (CHA), Munich
  - Universitäts-Kinderklinik Würzburg, Würzburg
- Ireland (5):
  - Cork University Hospital, Cork
  - Our Lady's Children's Hospital, Dublin
  - The National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Beaumont Hospital, Dublin
- United Kingdom (2):
  - Belfast City Hospital, Belfast, Northern Ireland
  - Imperial College London, London

REFERENCES:
- [Background] Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Drevinek P, Griese M, McKone EF, Wainwright CE, Konstan MW, Moss R, Ratjen F, Sermet-Gaudelus I, Rowe SM, Dong Q, Rodriguez S, Yen K, Ordonez C, Elborn JS; VX08-770-102 Study Group. A CFTR potentiator in patients with cystic fibrosis and the G551D mutation. N Engl J Med. 2011 Nov 3;365(18):1663-72. doi: 10.1056/NEJMoa1105185. PMID 22047557
- [Derived] Flume PA, Wainwright CE, Elizabeth Tullis D, Rodriguez S, Niknian M, Higgins M, Davies JC, Wagener JS. Recovery of lung function following a pulmonary exacerbation in patients with cystic fibrosis and the G551D-CFTR mutation treated with ivacaftor. J Cyst Fibros. 2018 Jan;17(1):83-88. doi: 10.1016/j.jcf.2017.06.002. Epub 2017 Jun 24. PMID 28651844
- [Derived] Solem CT, Vera-Llonch M, Liu S, Botteman M, Castiglione B. Impact of pulmonary exacerbations and lung function on generic health-related quality of life in patients with cystic fibrosis. Health Qual Life Outcomes. 2016 Apr 21;14:63. doi: 10.1186/s12955-016-0465-z. PMID 27097977
- [Derived] Quittner A, Suthoff E, Rendas-Baum R, Bayliss MS, Sermet-Gaudelus I, Castiglione B, Vera-Llonch M. Effect of ivacaftor treatment in patients with cystic fibrosis and the G551D-CFTR mutation: patient-reported outcomes in the STRIVE randomized, controlled trial. Health Qual Life Outcomes. 2015 Jul 2;13:93. doi: 10.1186/s12955-015-0293-6. PMID 26135562
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started on 10 June 2009 (signing of first informed consent). After obtaining consent and assent (where applicable), screening evaluations were completed during a period of 2 to 5 weeks (Day -35 to Day -15) before the first dose of study drug.
Pre-assignment Details: A total of 167 subjects were randomized; 161 subjects received at least 1 dose of the study drug. A 2-week run-in period was included to establish the baseline assessments on Day 1 after ensuring that subjects were properly taking their cystic fibrosis (CF) medication regimens.
Groups:
- Placebo: Oral tablet every 12 hours (q12h) for up to 48 weeks.
- 150 mg Ivacaftor q12h: Oral tablet of 150 mg of ivacaftor q12h for up to 48 weeks.
Period: Overall Study
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Started | 78 (All subjects who received at least 1 dose of study drug (placebo).) | 83 (All subjects who received at least 1 dose of study drug (ivacaftor).)
Completed Treatment Period, Week 24 | 71 | 80
Completed | 68 (Completed Treatment and Extension Periods (Through Week 48)) | 77 (Completed Treatment and Extension Periods (Through Week 48))
Not Completed | 10 | 6
Not completed — Adverse Event | 4 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Prohibited Medication | 2 | 1
Not completed — Withdrawal of Consent | 1 | 1
Not completed — Noncompliance with Study Requirements | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Wrong Genotype | 1 | 0
Not completed — Increased Lab Draws, Difficult Lab Stick | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 150 mg Ivacaftor q12h | Total
Number analyzed (Participants) | 78 | 83 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 19 | 36
  Between 18 and 65 years | 61 | 64 | 125
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.7 (9.21) | 26.2 (9.85) | 25.5 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 38 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 77 | 81 | 158
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 77 | 81 | 158
  Not Allowed to Ask Per Local Regulations | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  North America | 50 | 50 | 100
  Europe | 19 | 23 | 42
  Australia | 9 | 10 | 19
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1), Continuous [Mean (Standard Deviation); unit: percentage] — Percent predicted for age, gender, and height.
  percentage | 63.7 (16.83) | 63.5 (16.14) | 63.6 (16.43)
Percent Predicted FEV1, Categorical [Number; unit: participants] — Percent predicted for age, gender, and height.
  participants
    < 70% predicted FEV1 | 45 | 49 | 94
    ≥ 70% predicted FEV1 | 33 | 34 | 67
Weight [Mean (Standard Deviation); unit: kilograms] | 61.2 (13.93) | 61.7 (14.26) | 61.5 (14.06)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 21.9 (3.49) | 21.7 (3.65) | 21.8 (3.56)
Sweat Chloride [Mean (Standard Deviation); unit: millimoles per liter] | 100.1 (10.63) | 100.4 (10.00) | 100.2 (10.28)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Mean Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 24
Description: Spirometry (as measured by FEV1) is a standardized assessment to evaluate lung function that is the most widely used endpoint in cystic fibrosis studies.
Time Frame: baseline through 24 weeks
Population: All randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo) and had available assessments during the time frame.
Measure: Least Squares Mean (Standard Error); unit: percent of predicted volume (L)
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 78 | 83
percent of predicted volume (L) | -0.2 (0.7) | 10.4 (0.7)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; The primary analysis for the primary efficacy variable was based on a Mixed-Effects Model for Repeated Measures (MMRM). The model included absolute change from baseline in percent predicted forced expiratory volume in 1 second (FEV1) as the dependent variable, treatment (ivacaftor versus placebo) and visit (Day 15, Week 8, Week 16, and Week 24) as fixed effects, and subject as a random effect, with adjustment for the continuous baseline values of age and percent predicted FEV1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The primary and key secondary endpoints were analyzed using Hochberg's step-up procedure: test 1, primary (α=0.05); test 2, CFQ-R resp domain (Wk24) and sweat chloride (Wk24)(α=0.05); Denominator degrees of freedom were estimated using the Kenward-Roger approximation; Mean Difference (Final Values) = 10.6, 95% CI 2-sided [8.6 to 12.6], Standard Error of Mean 1.0

2. Secondary Outcome: Absolute Mean Change From Baseline in Percent Predicted FEV1 Through Week 48
Description: as for outcome 1
Time Frame: baseline through 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent of predicted volume (L)
Groups:
- 150 mg Ivacaftor q12h: Oral tablets of 150 mg of ivacaftor q12h for up to 48 weeks.
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 78 | 83
percent of predicted volume (L) | -0.4 (0.7) | 10.1 (0.7)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Analysis of this variable was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were obtained from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for the continuous baseline values of age and percent predicted forced expiratory volume in 1 second (FEV1),using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — There was no adjustment for multiple comparisons; Denominator degrees of freedom were estimated using the Kenward-Roger approximation. No imputation of missing data was done; Mean Difference (Final Values) = 10.5, 95% CI 2-sided [8.5 to 12.5], Standard Error of Mean 1.0

3. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Score Through Week 24 and Week 48 (Respiratory Domain Score, Pooled)
Description: The CFQ-R is a health-related quality of life measure for subjects with cystic fibrosis. Each domain is scored from 0 (worst) to 100 (best). A difference of at least 4 points in the respiratory domain score of the CFQ-R is considered a minimal clinically important difference (MCID).
Time Frame: baseline through 24 weeks and 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 71 | 80
score on a scale
  Change from Baseline Through Week 24 | -2.1 (1.3) | 6.0 (1.2)
  Change from Baseline Through Week 48 | -2.7 (1.2) | 6.0 (1.1)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 24: Analysis for the respiratory domain score endpoint was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous baseline value for age, domain score, and percent predicted FEV1, using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Analyzed in sequence: test 1, primary (α=0.05); test 2, using Hochberg's step-up procedure on CFQ-R resp domain(Wk 24) and sweat chloride (Wk 24) (α=0.05); Mean Difference (Final Values) = 8.1, 95% CI 2-sided [4.7 to 11.4], Standard Error of Mean 1.7
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 48: Analysis for the CFQ-R respiratory domain score endpoint was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from MMRM with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous baseline value for age,sweat chloride, and percent predicted FEV1,using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — There was no adjustment for multiple comparisons; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [5.3 to 11.9], Standard Error of Mean 1.7

4. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride Concentration Through Week 24 and Week 48
Description: The sweat chloride (quantitative pilocarpine iontophoresis) test is a standard diagnostic tool for cystic fibrosis (CF), serving as an indicator of cystic fibrosis transmembrane conductance regulator (CFTR) activity.
Time Frame: baseline through 24 weeks and 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 74 | 78
millimoles per liter
  Change from Baseline Through Week 24 | -0.8 (1.3) | -48.7 (1.2)
  Change from Baseline Through Week 48 | -0.6 (1.3) | -48.7 (1.2)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 24: Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous baseline value for age, sweat chloride, and percent predicted FEV1, using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Analyzed in sequence: test 1, primary (α=0.05); test 2, using Hochberg's step-up procedure on CFQ-R resp domain(Wk 24) and sweat chloride (Wk 24) (α=0.05); test 3 using Hochberg's on time to pulmonary exacerbation (Wk 48) and weight (Wk 48); Mean Difference (Final Values) = -47.9, 95% CI 2-sided [-51.3 to -44.5], Standard Error of Mean 1.7
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 48: Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous baseline value for age, sweat chloride, and percent predicted FEV1, using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — There was no adjustment for multiple comparisons; Mean Difference (Final Values) = -48.1, 95% CI 2-sided [-51.5 to -44.7], Standard Error of Mean 1.7

5. Secondary Outcome: Time-to-first Pulmonary Exacerbation Through Week 24 and Week 48
Description: Pulmonary exacerbation was defined as a change in antibiotic therapy (intravenous, inhaled, or oral) for any 4 or more of signs/symptoms such as change in sputum; new or increased hemoptysis; increased cough or dyspnea; malaise, fatigue, or lethargy; temperature above 38 degrees C; anorexia or weight loss; sinus pain/tenderness and discharge; change in physical examination of the chest; decreased pulmonary function by 10%; and radiographic changes indicative of pulmonary infection.
Time Frame: baseline through 24 weeks and 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of event-free participants
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 78 | 83
proportion of event-free participants
  0 to 15 Days | 0.97 [0.90 to 0.99] | 0.98 [0.91 to 0.99]
  16 to 56 Days | 0.87 [0.77 to 0.93] | 0.89 [0.80 to 0.94]
  57 to 112 Days | 0.72 [0.61 to 0.81] | 0.83 [0.73 to 0.90]
  113 to 168 Days | 0.53 [0.41 to 0.64] | 0.78 [0.68 to 0.86]
  169 to 224 Days | 0.51 [0.39 to 0.61] | 0.75 [0.64 to 0.83]
  225 to 280 Days | 0.44 [0.32 to 0.55] | 0.70 [0.58 to 0.78]
  281 to 336 Days | 0.41 [0.29 to 0.52] | 0.67 [0.55 to 0.76]
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Time to first pulmonary exacerbation through Week 24 was analyzed using Cox regression. The model included a covariate for treatment and adjustments for the age group and percent predicted forced expiratory volume in 1 second (FEV1) severity at baseline; Test type: Superiority or Other; p = 0.0016, Regression, Cox — There was no adjustment for multiple comparisons; Cox Proportional Hazard at Week 24 = 0.40, 95% CI 2-sided [0.23 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; Time to first pulmonary exacerbation through Week 48 was analyzed using Cox regression. The model included a covariate for treatment and adjustments for the age group and percent predicted forced expiratory volume in 1 second (FEV1) severity at baseline; Test type: Superiority or Other; p = 0.0012, Regression, Cox — [p-value comment as in outcome 4, analysis 1]; Cox Proportional Hazard at 48 Weeks = 0.46, 95% CI 2-sided [0.28 to 0.73]

6. Secondary Outcome: Absolute Change From Baseline in Weight at Week 24 and Week 48
Description: As malnutrition is common in patients with cystic fibrosis (CF) because of increased energy expenditures due to lung disease and fat malabsorption, body weight is an important clinical measure of nutritional status.
Time Frame: baseline to 24 weeks and 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 78 | 83
kilograms
  At Week 24 | 0.2 (0.4) | 3.0 (0.4)
  At Week 48 | 0.4 (0.5) | 3.1 (0.5)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; At Week 24: Analysis for this variable was based on a linear mixed effects (LME) model with treatment as a fixed effect, and intercept, visit (days on study) and treatment by visit interaction as random effects, with adjustment for age group and baseline percent predicted forced expiratory volume in 1 second (FEV1) severity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; There was no adjustment for multiple comparisons; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [1.8 to 3.7], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; At Week 48: Analysis for this variable was based on a linear mixed effects (LME) model with treatment as a fixed effect and visit (days on study) and treatment by visit interaction as random effects, with adjustment for age group and baseline percent predicted forced expiratory volume in 1 second (FEV1) severity; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [1.3 to 4.1], Standard Error of Mean 0.7

ADVERSE EVENTS:
Time Frame: For enrolled subjects, adverse events were collected through the Follow-up Visit (4 weeks [± 7 days] after the last dose of study drug).
Description: For subjects who were screened but were not subsequently enrolled in the study, non-serious AEs were not collected, but SAEs were reported. For subjects who completed 48 weeks of study drug treatment and enrolled in the open-label extension study, adverse events were only collected through the Week 48 Visit.
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Serious Adverse Events (participants affected / at risk) | 33/78 | 20/83
Other Adverse Events (participants affected / at risk) | 78/78 | 82/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | 150 mg Ivacaftor q12h (N=83)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 26 (37) | 11 (22) — CF exacerbations were coded as "cystic fibrosis lung."
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter related complication (General disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Myringitis bullous (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | 150 mg Ivacaftor q12h (N=83)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (59) | 27 (38)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (23) | 17 (25)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 17 (22)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 9 (17)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (19) | 12 (15)
Rales (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 9 (17)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (7)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 12 (16) | 19 (26)
Nasopharyngitis (Infections and infestations) | 10 (14) | 10 (13)
Sinusitis (Infections and infestations) | 7 (12) | 6 (8)
Rhinitis (Infections and infestations) | 4 (4) | 6 (6)
Viral infection (Infections and infestations) | 5 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (13) | 13 (14)
Nausea (Gastrointestinal disorders) | 9 (12) | 13 (22)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 11 (12)
Vomiting (Gastrointestinal disorders) | 10 (10) | 9 (13)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 4 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Pulmonary function test decreased (Investigations) | 11 (14) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (6) | 5 (9)
C-reactive protein increased (Investigations) | 5 (6) | 4 (4)
Blood glucose increased (Investigations) | 3 (3) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (7)
Bacteria sputum identified (Investigations) | 1 (1) | 6 (7)
Breath sounds abnormal (Investigations) | 4 (5) | 2 (2)
Weight decreased (Investigations) | 4 (4) | 2 (2)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 39 (77) | 29 (47) — CF exacerbations were coded as "cystic fibrosis lung."
Headache (Nervous system disorders) | 13 (31) | 19 (39)
Dizziness (Nervous system disorders) | 1 (1) | 10 (11)
Sinus headache (Nervous system disorders) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 12 (22)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Pyrexia (General disorders) | 9 (11) | 10 (13)
Fatigue (General disorders) | 7 (9) | 7 (8)
Joint sprain (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days